CLINICAL TRIAL: NCT02662517
Title: Growth Hormones and Cells in Human Milk Depending on Gestational Age and Lactation Phase
Brief Title: Growth Hormones and Cells in Human Milk Depending on Gestational Age
Acronym: BMProfile
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Titus Keller, MD, Neonatologist, University Hospital of Cologne
Other Study IDs: UHCologne
Record Dates: First submitted 2016-01-11; First posted 2016-01-25 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Lactation
Keywords: Neurotrophins; Stem Cells; Prematurity
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human breast milk, umbilical chord blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Human breast milk contains growth factors including neurotrophins and cells with neuroprotective potential. Concerning growth factors milk of preterms differs significantly from term milk. The aim of this study is to give a profile of human milk concerning non-nutritive factors depending on gestational age and lactation phase.

DETAILED DESCRIPTION:
Neurotrophins (epidermal growth factor (EGF), vascular endothelial growth factor (VEGF), nerve growth factor (NGF), brain derived neurotrophic factor (BDNF)) as well as amount of cells, especially positive for sex-determining transformer protein (TRA)-1-81 and stage-specific embryonic antigen (SSEA)-4, are planned to be quantified in human breast milk of extremely preterm newborns as well as term newborns at different stages of lactation.

ELIGIBILITY:
Inclusion Criteria:

* the newborn infant is being fed with own mothers milk

Exclusion Criteria:

* low amount of breast milk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breastfeeding mothers
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-03-01; Primary Completion 2016-09-30 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
neurotrophins composition | day 7
  Concentration of Neurotrophins EGF, VEGF, NGF, BDNF in the human milk

SECONDARY OUTCOMES:
Amount of cells positive for surface markers TRA-1-81 and SSEA-4 | day 7
  surface markers characteristic for pluripotent stem cells

CONTACTS AND LOCATIONS:
Overall Officials: Titus Keller, MD, Principal Investigator — Neonatology, University Hospital of Cologne
Locations (1):
- Neonatology at the University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Keller T, Wengenroth L, Smorra D, Probst K, Kurian L, Kribs A, Brachvogel B. Novel DRAQ5/SYTOX(R) Blue Based Flow Cytometric Strategy to Identify and Characterize Stem Cells in Human Breast Milk. Cytometry B Clin Cytom. 2019 Nov;96(6):480-489. doi: 10.1002/cyto.b.21748. Epub 2018 Nov 26. PMID 30479054